CLINICAL TRIAL: NCT03291379
Title: VEROnA: A Window of Opportunity Study of Vandetanib-eluting Radiopaque Embolic Beads (BTG-002814) in Patients With Resectable Liver Malignancies
Brief Title: Vandetanib-eluting Radiopaque Embolic Beads in Patients With Resectable Liver Malignancies
Acronym: VEROnA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTG-002814-01
Record Dates: First submitted 2017-05-17; First posted 2017-09-25 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Carcinoma, Hepatocellular; Metastatic Colorectal Cancer
Keywords: mCRC, HCC, radiopaque beads, vandetanib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: 1 mL BTG-002814 containing 100 mg vandetanib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BTG-002814 (Experimental): Single arm: BTG-002814 (vandetanib-eluting radiopaque beads)
  Interventions: Drug: BTG-002814

INTERVENTIONS:
Drug: BTG-002814 — BTG-002814 containing 100 mg vandetanib
  Other Names: vandetanib-eluting radiopaque beads

SUMMARY:
This is a pilot, open label single arm phase 0 window of opportunity study of vandetanib-eluting radiopaque beads in patients with resectable liver malignancies.

DETAILED DESCRIPTION:
A pilot open-label single arm multicenter phase 0 window of opportunity study of BTG-002814 given up to 3 weeks prior to surgery in up to 12 patients with resectable Hepatocellular carcinoma (HCC) or Colorectal cancer (CRC) with liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults (≥ 18 years old)
2. Patient with resectable HCC (Child Pugh A, International Normalized Ratio (INR) ≤1.5) or resectable liver metastases from CRC and a candidate for liver surgery
3. Patients with low risk for surgical morbidity and mortality from liver surgery according to the investigators judgement
4. World Health Organization (WHO) performance status 0, 1 or 2
5. Adequate haematological function with Hb >90 g/L, absolute neutrophil count >1.5 x 10^9/L, Plt >100 x 10^9/L
6. Adequate liver function with serum bilirubin <1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) (or aspartate aminotransferase (AST) if ALT not available) ≤5 x ULN, alkaline phosphatase (ALP) <5 x ULN
7. Adequate renal function with serum creatinine ≤1.5 x ULN and calculated creatinine clearance (GFR) ≥50 mL/min estimated using a validated creatinine clearance calculation (e.g., Cockcroft-Gault or Wright formula).
8. Patient is willing to provide blood samples, and tissue samples at surgical resection, for research purposes
9. Patient is willing and able to provide written informed consent

Exclusion Criteria:

1. Any systemic chemotherapy within 3 months of the screening visit or any plan to administer systemic chemotherapy prior to surgery
2. Previous treatment with transarterial embolisation (with or without chemotherapy) of the liver, prior radiotherapy or ablation therapy to the liver or prior yttrium-90 microsphere therapy
3. Any contraindication to vandetanib according to its local label including:

   * Hypersensitivity to the active substance
   * Congenital long corrected QT interval (QTc) syndrome
   * Patients known to have a QTc interval over 480 milliseconds
   * Concomitant use of medicinal products known to also prolong the QTc interval and/or induce Torsades de pointes
4. Any contraindication to hepatic artery catheterisation or hepatic embolisation procedures (e.g. portal venous thrombosis, severely reduced portal venous flow or hepatofugal blood flow, untreated varices at high risk of bleeding)
5. Women of childbearing potential not using effective contraception or women who are breast feeding
6. Confirmed allergy to iodine-based intravenous contrast media
7. Patients who cannot have CT, MRI or dynamic contrast-enhanced (DCE) MRI Imaging (according to site policy)
8. Active uncontrolled cardiovascular disease
9. Any co-morbid disease or condition or event that, in the investigator's judgment, would place the patient at undue risk and would preclude the safe use of BTG-002814
10. Levels of potassium, calcium, magnesium or thyroid stimulating hormone (TSH) outside the normal ranges, and that in the investigator's judgement are clinically significant, or other laboratory findings that in the view of the investigator makes it undesirable for the patient to participate in the study
11. Patients who have participated in another clinical trial with an investigational product within 4 weeks prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2019-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ricky Sharma, Principal Investigator — University College, London
Locations (1):
- University College London Hospital, Bloomsbury, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beaton L, Tregidgo HFJ, Znati SA, Forsyth S, Clarkson MJ, Bandula S, Chouhan M, Lowe HL, Zaw Thin M, Hague J, Sharma D, Pollok JM, Davidson BR, Raja J, Munneke G, Stuckey DJ, Bascal ZA, Wilde PE, Cooper S, Ryan S, Czuczman P, Boucher E, Hartley JA, Lewis AL, Jansen M, Meyer T, Sharma RA. VEROnA Protocol: A Pilot, Open-Label, Single-Arm, Phase 0, Window-of-Opportunity Study of Vandetanib-Eluting Radiopaque Embolic Beads (BTG-002814) in Patients With Resectable Liver Malignancies. JMIR Res Protoc. 2019 Oct 2;8(10):e13696. doi: 10.2196/13696. PMID 31579027

RESULTS

PARTICIPANT FLOW:
Groups:
- BTG-002814: Single arm: BTG-002814 (vandetanib-eluting radiopaque beads)
  BTG-002814 (vandetanib-eluting radiopaque beads): BTG-002814 containing 100 mg vandetanib
Period: Overall Study
Arm/Group | BTG-002814
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BTG-002814
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 62.5 [50 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8
World Health Organisation (WHO) Performance Status [Count of Participants; unit: Participants]
  Grade 0 (asymptomatic) | 8
  Grade 1 (Symptomatic, but ambulatory) | 0
  Grade 2 (Symptomatic, <50% in bed) | 0
Tumour type [Count of Participants; unit: Participants] — Participants must have resectable Hepatocellular carcinoma (HCC) (Child Pugh A, international normalized ratio (INR) ≤1.5) or resectable liver metastases from colorectal cancer (CRC) and be a candidate for liver surgery
  Participants
    Hepatocellular carcinoma (HCC) | 2
    Metastatic colorectal cancer (mCRC) | 6
Number of liver lesions [Mean (Standard Deviation); unit: Count] | 1.6 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Safety and Tolerability of Treatment With BTG-002814
Description: Adverse events (AEs) related to treatment with BTG-002814 using the National Cancer Institute- Common Terminology Criteria for Adverse Events- Version 4.0 (NCI-CTCAE v4.0)
Time Frame: Continuously throughout the study totalling 9 weeks
Population: Safety population - all participants treated with BTG-002814
Measure: Count of Participants; unit: Participants
Arm/Group | BTG-002814
Number analyzed (Participants) | 8
Participants
  participants with treatment emergent Adverse Events (AEs) | 8
  participants with treatment emergent Serious Adverse Events (SAEs) | 4

2. Primary Outcome: Maximum Concentration (Cmax) of Vandetanib and N-desmethyl Vandetanib in Plasma Following Treatment With BTG-002814
Description: Pharmacokinetic (PK) analysis of participants plasma samples by liquid chromatography with tandem mass spectrometry at the following timepoints: pre-treatment, post treatment (2 hours, 4 hours, 24 hours), prior to surgery, and end of study to derive Cmax.
Time Frame: pre-treatment, 2 hours post-treatment, 4 hours post treatment, 24 hours post treatment, prior to surgery, and end of study (28-32 days post-surgery)
Population: all participants treated with BTG-002814
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BTG-002814
Number analyzed (Participants) | 8
ng/mL
  Vandetanib Plasma Cmax | 24.3 (13.94)
  N-desmethyl Plasma Cmax | 0.6 (0.82)

3. Primary Outcome: Concentration of Vandetanib in Resected Liver Tissue Following Treatment With BTG-002814
Description: PK analysis of participants resected liver tissue samples by liquid chromatography with tandem mass spectrometry to determine vandetanib concentrations at the centre, middle, and edge of the tumour, as well as in the normal tissue surrounding the tumour (1cm away).
Time Frame: Following surgical resection of tumour
Population: Results were not available for 2 patients where sample was incorrectly prepared, or no sample was received. For patients with multiple tumours, only the treated tumours were sampled and analysed. The results for this outcome measure are reported by individual subject (where data was available) by each sample location (centre, middle, edge of the tumour or 1cm away from tumour) per row.
Measure: Number; unit: ng/mL
Arm/Group | BTG-002814
Number analyzed (Participants) | 6
ng/mL
  Subject 01: Vandetanib concentration centre of tumour: number analyzed (Participants) | 1
  Subject 01: Vandetanib concentration centre of tumour | 404000
  Subject 01: Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 01: Vandetanib concentration middle of tumour | 394000
  Subject 01: Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 01: Vandetanib concentration edge of tumour | 327000
  Subject 01: Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 01: Vandetanib concentration 1cm away from tumour | 10800
  Subject 03: Vandetanib concentration centre of tumour: number analyzed (Participants) | 1
  Subject 03: Vandetanib concentration centre of tumour | 8510
  Subject 03: Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 03: Vandetanib concentration middle of tumour | 11000
  Subject 03: Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 03: Vandetanib concentration edge of tumour | 18800
  Subject 03: Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 03: Vandetanib concentration 1cm away from tumour | 9120
  Subject 05: Vandetanib concentration centre of tumour: number analyzed (Participants) | 1
  Subject 05: Vandetanib concentration centre of tumour | 7340
  Subject 05: Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 05: Vandetanib concentration middle of tumour | 7550
  Subject 05: Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 05: Vandetanib concentration edge of tumour | 12500
  Subject 05: Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 05: Vandetanib concentration 1cm away from tumour | 7090
  Subject 06: Vandetanib concentration centre of tumour: number analyzed (Participants) | 1
  Subject 06: Vandetanib concentration centre of tumour | 160000
  Subject 06: Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 06: Vandetanib concentration middle of tumour | 151000
  Subject 06: Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 06: Vandetanib concentration edge of tumour | 11100
  Subject 06: Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 06: Vandetanib concentration 1cm away from tumour | 1480
  Subject 07: Vandetanib concentration centre of tumour: number analyzed (Participants) | 1
  Subject 07: Vandetanib concentration centre of tumour | 4570
  Subject 07: Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 07: Vandetanib concentration middle of tumour | 531
  Subject 07: Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 07: Vandetanib concentration edge of tumour | 441
  Subject 07: Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 07: Vandetanib concentration 1cm away from tumour | 2760
  Subject 08: Vandetanib concentration centre of tumour: number analyzed (Participants) | 1
  Subject 08: Vandetanib concentration centre of tumour | 1140
  Subject 08 (1cm lesion): whole tumour Vandetanib concentration: number analyzed (Participants) | 1
  Subject 08 (1cm lesion): whole tumour Vandetanib concentration | 93500
  Subject 08 (inferior lesion): Vandetanib concentration centre of tumour: number analyzed (Participants) | 1
  Subject 08 (inferior lesion): Vandetanib concentration centre of tumour | 6180
  Subject 08: Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 08: Vandetanib concentration middle of tumour | 1240
  Subject 08 (inferior lesion): Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 08 (inferior lesion): Vandetanib concentration middle of tumour | 1440
  Subject 08: Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 08: Vandetanib concentration edge of tumour | 2840
  Subject 08 (inferior lesion): Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 08 (inferior lesion): Vandetanib concentration edge of tumour | 2710
  Subject 08: Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 08: Vandetanib concentration 1cm away from tumour | 29100
  Subject 08 (1 cm lesion): Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 08 (1 cm lesion): Vandetanib concentration 1cm away from tumour | 5350
  Subject 08 (inferior lesion): Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 08 (inferior lesion): Vandetanib concentration 1cm away from tumour | 6010

4. Primary Outcome: Time Taken to Reach the Maximum Concentration (Tmax) of Vandetanib and N-desmethyl Vandetanib in Plasma Following Treatment With BTG-002814
Description: PK analysis of participants plasma samples by liquid chromatography with tandem mass spectrometry at the following timepoints: pre-treatment, post treatment (2 hours, 4 hours, 24 hours), prior to surgery, and end of study to derive Tmax
Time Frame: as for outcome 2
Population: all participants treated with BTG-002814
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BTG-002814
Number analyzed (Participants) | 8
hours
  Vandetanib Plasma Tmax | 26.0 (67.08)
  N-desmethyl Plasma Tmax | 0.8 (1.04)

5. Primary Outcome: Concentration of Vandetanib and N-desmethyl Vandetanib in Plasma Over Time Until End of Study Following Treatment With BTG-002814
Description: PK analysis of participants plasma samples by liquid chromatography with tandem mass spectrometry at the following timepoints: pre-treatment, post treatment (2 hours, 4 hours, 24 hours), prior to surgery, and end of study to derive AUCEoS (area under the curve at end of study).
Time Frame: as for outcome 2
Population: all participants treated with BTG-002814
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | BTG-002814
Number analyzed (Participants) | 8
ng*h/mL
  Vandetanib Plasma AUCEoS | 6979.3 (3188.21)
  N-desmethyl Plasma AUCEoS | 81.1 (169.40)

6. Primary Outcome: Concentration of N-desmethyl Vandetanib in Resected Liver Tissue Following Treatment With BTG-002814
Description: PK analysis of participants resected liver tissue samples by liquid chromatography with tandem mass spectrometry to determine N-desmethyl vandetanib concentrations at the centre, middle, and edge of the tumour, as well as in the normal tissue surrounding the tumour (1cm away).
Time Frame: Following surgical resection of tumour
Population: Results were not available for 2 patients where sample was incorrectly prepared, or no sample was received. For patients with multiple tumours, only the treated tumours were sampled and analysed. The results for this outcome measure are reported by individual subject (where data was available), by each sample location (centre, middle, edge of the tumour, 1cm away from tumour) per row.
Measure: Number; unit: ng/mL
Arm/Group | BTG-002814
Number analyzed (Participants) | 6
ng/mL
  Subject 01: N-desmethyl Vandetanib concentration centre of tumour: number analyzed (Participants) | 1
  Subject 01: N-desmethyl Vandetanib concentration centre of tumour | 4620
  Subject 01: N-desmethyl Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 01: N-desmethyl Vandetanib concentration middle of tumour | 4740
  Subject 01: N-desmethyl Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 01: N-desmethyl Vandetanib concentration edge of tumour | 3680
  Subject 01: N-desmethyl Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 01: N-desmethyl Vandetanib concentration 1cm away from tumour | 280
  Subject 03: N-desmethyl concentration centre of tumour: number analyzed (Participants) | 1
  Subject 03: N-desmethyl concentration centre of tumour | 69.6
  Subject 03: N-desmethyl Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 03: N-desmethyl Vandetanib concentration middle of tumour | 59.8
  Subject 03: N-desmethyl Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 03: N-desmethyl Vandetanib concentration edge of tumour | 69.2
  Subject 03: N-desmethyl Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 03: N-desmethyl Vandetanib concentration 1cm away from tumour | 831
  Subject 05: N-desmethyl concentration centre of tumour: number analyzed (Participants) | 1
  Subject 05: N-desmethyl concentration centre of tumour | 421
  Subject 05: N-desmethyl Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 05: N-desmethyl Vandetanib concentration middle of tumour | 418
  Subject 05: N-desmethyl Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 05: N-desmethyl Vandetanib concentration edge of tumour | 469
  Subject 05: N-desmethyl Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 05: N-desmethyl Vandetanib concentration 1cm away from tumour | 544
  Subject 06: N-desmethyl concentration centre of tumour: number analyzed (Participants) | 1
  Subject 06: N-desmethyl concentration centre of tumour | 113
  Subject 06: N-desmethyl Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 06: N-desmethyl Vandetanib concentration middle of tumour | 93.9
  Subject 06: N-desmethyl Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 06: N-desmethyl Vandetanib concentration edge of tumour | 11.4
  Subject 06: N-desmethyl Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 06: N-desmethyl Vandetanib concentration 1cm away from tumour | 55.6
  Subject 07: N-desmethyl concentration centre of tumour: number analyzed (Participants) | 1
  Subject 07: N-desmethyl concentration centre of tumour | 21
  Subject 07: N-desmethyl Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 07: N-desmethyl Vandetanib concentration middle of tumour | 15.7
  Subject 07: N-desmethyl Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 07: N-desmethyl Vandetanib concentration edge of tumour | 28.7
  Subject 07: N-desmethyl Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 07: N-desmethyl Vandetanib concentration 1cm away from tumour | 84
  Subject 08: N-desmethyl concentration centre of tumour: number analyzed (Participants) | 1
  Subject 08: N-desmethyl concentration centre of tumour | 39.3
  Subject 08 (1cm lesion): whole tumour N-desmethyl concentration: number analyzed (Participants) | 1
  Subject 08 (1cm lesion): whole tumour N-desmethyl concentration | 208
  Subject 08 (inferior lesion): N-desmethyl concentration centre of tumour: number analyzed (Participants) | 1
  Subject 08 (inferior lesion): N-desmethyl concentration centre of tumour | 80.2
  Subject 08: N-desmethyl Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 08: N-desmethyl Vandetanib concentration middle of tumour | 57.1
  Subject 08 (inferior lesion): N-desmethyl Vandetanib concentration middle of tumour: number analyzed (Participants) | 1
  Subject 08 (inferior lesion): N-desmethyl Vandetanib concentration middle of tumour | 101
  Subject 08: N-desmethyl Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 08: N-desmethyl Vandetanib concentration edge of tumour | 145
  Subject 08 (inferior lesion): N-desmethyl Vandetanib concentration edge of tumour: number analyzed (Participants) | 1
  Subject 08 (inferior lesion): N-desmethyl Vandetanib concentration edge of tumour | 171
  Subject 08: N-desmethyl Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 08: N-desmethyl Vandetanib concentration 1cm away from tumour | 389
  Subject 08 (1 cm lesion): N-desmethyl Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 08 (1 cm lesion): N-desmethyl Vandetanib concentration 1cm away from tumour | 342
  Subject 08 (inferior lesion): N-desmethyl Vandetanib concentration 1cm away from tumour: number analyzed (Participants) | 1
  Subject 08 (inferior lesion): N-desmethyl Vandetanib concentration 1cm away from tumour | 405

7. Secondary Outcome: Evaluate the Anatomical Distribution of BTG-002814 on Non-contrast Enhanced Imaging Using 4D CT
Description: An automated thresholding and filtering algorithm was designed to allow the volume of delivered beads to be quantitatively determined for regions of interest (liver, registered sample, tumour, tumour dilated 1cm, tumour dilated 2cm) from the pre-surgical non-contrast CT scan and the PET/CT of the explanted liver samples following surgery.
Time Frame: 1 day after treatment
Population: All 8 subjects treated with BTG-002814 were analysed, however, not all subjects have sampling of all regions (liver, registered sample, tumour, tumour dilated 1cm, tumour dilated 2cm) due to some samples not being able to be accurately processed and registered. The data for this outcome measure is reported by individual subject, for each sample region (where data is available) per row.
Measure: Number; unit: µL
Arm/Group | BTG-002814
Number analyzed (Participants) | 8
µL
  Subject 01: Liver: number analyzed (Participants) | 1
  Subject 01: Liver | 928.83
  Subject 01: Registered sample: number analyzed (Participants) | 1
  Subject 01: Registered sample | 399.27
  Subject 01: Tumour: number analyzed (Participants) | 1
  Subject 01: Tumour | 361.14
  Subject 01: tumour dilated 1cm: number analyzed (Participants) | 1
  Subject 01: tumour dilated 1cm | 393.79
  Subject 01: Tumour dilated 2cm: number analyzed (Participants) | 1
  Subject 01: Tumour dilated 2cm | 479.28
  Subject 02: Liver: number analyzed (Participants) | 1
  Subject 02: Liver | 764.69
  Subject 02: Tumour: number analyzed (Participants) | 1
  Subject 02: Tumour | 596.78
  Subject 02: Tumour dilated 1cm: number analyzed (Participants) | 1
  Subject 02: Tumour dilated 1cm | 617.72
  Subject 02: Tumour dilated 2cm: number analyzed (Participants) | 1
  Subject 02: Tumour dilated 2cm | 649.97
  Subject 03: Liver: number analyzed (Participants) | 1
  Subject 03: Liver | 594.79
  Subject 03: Registered sample: number analyzed (Participants) | 1
  Subject 03: Registered sample | 116.54
  Subject 03: Tumour: number analyzed (Participants) | 1
  Subject 03: Tumour | 0.32
  Subject 03: Tumour dilated 1cm: number analyzed (Participants) | 1
  Subject 03: Tumour dilated 1cm | 36.26
  Subject 03: Tumour dilated 2cm: number analyzed (Participants) | 1
  Subject 03: Tumour dilated 2cm | 108.85
  Subject 04: Liver: number analyzed (Participants) | 1
  Subject 04: Liver | 852.03
  Subject 05: Liver: number analyzed (Participants) | 1
  Subject 05: Liver | 849.29
  Subject 05: Registered sample: number analyzed (Participants) | 1
  Subject 05: Registered sample | 751.62
  Subject 05: Tumour: number analyzed (Participants) | 1
  Subject 05: Tumour | 0
  Subject 5: Tumour dilated 1cm: number analyzed (Participants) | 1
  Subject 5: Tumour dilated 1cm | 15.26
  Subject 05: Tumour dilated 2cm: number analyzed (Participants) | 1
  Subject 05: Tumour dilated 2cm | 86.28
  Subject 06: Liver: number analyzed (Participants) | 1
  Subject 06: Liver | 202.56
  Subject 06: Registered sample: number analyzed (Participants) | 1
  Subject 06: Registered sample | 148.09
  Subject 06: Tumour: number analyzed (Participants) | 1
  Subject 06: Tumour | 51.14
  ubject 06: Tumour dilated 1cm: number analyzed (Participants) | 1
  ubject 06: Tumour dilated 1cm | 115.39
  Subject 06: Tumour dilated 2cm: number analyzed (Participants) | 1
  Subject 06: Tumour dilated 2cm | 166.80
  Subject 07: Liver: number analyzed (Participants) | 1
  Subject 07: Liver | 720.78
  Subject 07: Registered sample: number analyzed (Participants) | 1
  Subject 07: Registered sample | 103.82
  Subject 07: Tumour: number analyzed (Participants) | 1
  Subject 07: Tumour | 4.32
  Subject 07: Tumour dilated 1cm: number analyzed (Participants) | 1
  Subject 07: Tumour dilated 1cm | 75.43
  Subject 07: Tumour dilated 2cm: number analyzed (Participants) | 1
  Subject 07: Tumour dilated 2cm | 133.26
  Subject 08: Liver: number analyzed (Participants) | 1
  Subject 08: Liver | 693.73
  Subject 08: Registered sample: number analyzed (Participants) | 1
  Subject 08: Registered sample | 422.37
  Subject 08: Tumour: number analyzed (Participants) | 1
  Subject 08: Tumour | 21.87
  Subject 08: Tumour dilated 1cm: number analyzed (Participants) | 1
  Subject 08: Tumour dilated 1cm | 264.90
  Subject 08: Tumour dilated 2cm: number analyzed (Participants) | 1
  Subject 08: Tumour dilated 2cm | 378.15

8. Secondary Outcome: Evaluation of Histopathological Features in the Surgical Specimen (Malignant and Non-malignant Liver Tissue) by Analysing Percentage of Tumour Necrosis and Viability
Description: An evaluation of histopathological features in both malignant and non-malignant liver tissue from the surgical specimen was performed by microscopic examination. Sections of resected liver tissue was paraffin-embedded and Hematoxylin and Eosin (H&E) slides were produced. The H&E slides were scanned to produce 3D pathology models of tumour volume and compared to the 3D models generated from clinical imaging. This allowed the extent of tumour necrosis and viable tumour to be determined.
Time Frame: Post-surgery (tumour resection)
Population: all participants treated with BTG-002814
Measure: Median (Full Range); unit: percentage of surgical specimen
Arm/Group | BTG-002814
Number analyzed (Participants) | 8
percentage of surgical specimen
  Tumour necrosis | 92.5 [5 to 100]
  Viable tumour | 7.5 [0 to 95]

9. Secondary Outcome: Evaluation of Histopathological Features in the Surgical Specimen (Malignant and Non-malignant Liver Tissue) by Assessing Number of Participants With Any Vascular Changes.
Description: An evaluation of histopathological features in both malignant and non-malignant liver tissue from the surgical specimen was performed by microscopic examination. Sections of resected liver tissue was paraffin-embedded and Hematoxylin and Eosin (H&E) slides were produced. The H&E slides were scanned to produce 3D pathology models of tumour volume and compared to the 3D models generated from clinical imaging. This allowed any vascular changes to be determined.
Time Frame: Post-surgery (tumour resection)
Measure: Number; unit: Count of Participants
Arm/Group | BTG-002814
Number analyzed (Participants) | 8
Count of Participants
  Vascular changes absent | 8
  Vascular changes present | 0

10. Secondary Outcome: Assessment of Changes in Blood Flow on Dynamic Contrast-Enhanced (DCE) MRI Following Treatment With BTG-002814. The Following Parameters Will be Derived From DCE-MRI Images: Ktrans, Kep and Ve.
Description: After acquisition of DCE-MRI liver sequences, tumour signal intensity curves were used to calculate tissue parameters describing tumour perfusion, blood flow and vascularity, before and following treatment with BTG 002814.
  Bland Altman analysis showed the variability between baseline and pre-treatment readings to be too high, so an interpretation of the changes in blood flow prior to surgery is unreliable.
Time Frame: Baseline, pre-treatment, up to 3 days prior to surgical resection of tumour
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Study Blood Biomarkers With the Potential to Identify Patients Likely to Respond to Treatment With BTG-002814
Description: The following serum biomarkers were measured at Baseline, pre-treatment, 1 day after treatment, Up to 3 days prior to surgical resection, end of study ; cytokines, chemokines and growth factors relevant to cancer and inflammation.
Time Frame: Baseline, pre-treatment, 1 day after treatment, Up to 3 days prior to surgical resection, end of study (28-32 days post-surgery).
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Study Tissue Biomarkers to Explore Key Immune, Inflammatory and Drug Related Mechanisms
Description: The following tissue biomarkers were measured at Baseline, pre-treatment, Up to 3 days prior to surgical resection; Levels of serum alpha-fetoprotein (AFP) in patients with HCC. Levels of serum Carcinoembryonic Antigen (CEA), Cancer Antigen (CA)19-9 and CA-125 in patients with metastatic colorectal cancer (mCRC).
Time Frame: Baseline, pre-treatment, Up to 3 days prior to surgical resection.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From date participant signed Informed Consent until the patient's last visit (up to 9 weeks) (or after this date if the site Investigator feels the event is related to study treatment)
Arm/Group | BTG-002814
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTG-002814 (N=8)
Ileus (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Ascites (Hepatobiliary disorders) | 1 (1)
Post procedural bile leak (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTG-002814 (N=8)
Bradycardia (Cardiac disorders) | 3 (5)
Cardiac signs and symptoms NEC (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (19)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (8)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (8)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 7 (23)
Influenza like illness (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (3)
Alanine aminotransferase (Investigations) | 5 (8)
Aspartate aminotransferase (Investigations) | 5 (7)
Blood albumin (Investigations) | 3 (25)
Blood alkaline phosphatase (Investigations) | 5 (5)
Blood bilirubin (Investigations) | 1 (1)
Blood calcium (Investigations) | 2 (2)
Blood creatinine (Investigations) | 2 (7)
Blood glucose (Investigations) | 5 (8)
Blood lactic acid (Investigations) | 1 (1)
Blood magnesium (Investigations) | 1 (1)
Blood sodium (Investigations) | 1 (1)
Blood thyroid stimulating hormone (Investigations) | 2 (2)
Blood urea (Investigations) | 2 (2)
Blood uric acid (Investigations) | 4 (6)
C-reactive protein (Investigations) | 1 (14)
Electrocardiogram QT prolonged (Investigations) | 2 (4)
Gamma-glutamyl transferase (Investigations) | 5 (8)
Glomerular filtration rate (Investigations) | 1 (1)
Haemoglobin (Investigations) | 8 (15)
International normalized ratio (Investigations) | 1 (1)
Neutrophil count (Investigations) | 1 (11)
Neutrophil count decreased (Investigations) | 4 (6)
Platelet count (Investigations) | 2 (2)
Weight decreased (Investigations) | 3 (3)
White blood cell count (Investigations) | 2 (14)
Decreased appetite (Metabolism and nutrition disorders) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 7 (12)
Hypotension (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT03291379/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT03291379/SAP_000.pdf